CLINICAL TRIAL: NCT04964635
Title: TETRAGRIP II - Usability Trial of an FES Orthosis for People With Tetraplegia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: Salisbury NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RED 10356
Record Dates: First submitted 2021-06-23; First posted 2021-07-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TetraGrip II system — This main aim of this whole research project is to evaluate the performance of the TetraGrip II system in improving the upper limb functions in people with C4-C7 tetraplegia i.e. people who have damaged their spinal cord in the neck resulting in loss of function in all four limbs. The Tetragrip system uses a technique called Functional Electrical Stimulation (FES) in which small electrical impulses are used to activate paralysed muscles and hence provide movement. The stimulation is controlled by sensors which measure the movement of the other shoulder and enable the person to regain the use of their hand via stimulating electrodes placed on the skin over the relevant muscles.
  The feasibility of using this FES based system in restoring the upper arm functions will be evaluated by clinically trying the device on participants with C4-C7 tetraplegia.

SUMMARY:
Functional Electrical Stimulation is an established technique in which small electrical impulses are used to cause a contraction in muscles and thereby enable movement, in people with neurological or musculoskeletal problems who are unable to undertake those movements themselves. People with spinal cord injuries of the neck at C5, C6 and C7 account for 35% of all spinal cord injuries. Despite this, there is only one commercial FES (Functional Electrical Stimulation) based orthosis currently available. Even that has limitations in that it as it has a single size rigid exoskeleton it does not fit all people who could benefit and also due to its rigidity it does not allow people with lower injuries to utilise any remaining tenodesis grip. As a result, it is not widely used within the spinal injured communities. Therefore what is required is a more flexible system that can benefit a larger number of people whilst still being affordable within the constraints of the NHS. A previous INSPIRE funded project, TETRAGRIP I demonstrated that a surface FES system controlled by an inertial sensor, measuring movement of the opposite shoulder, could meet this specification and was successfully tried on two people with tetraplegia. What is now required is a more detailed study in which the principle components of that system are incorporated into a practical device suitable for use at home without clinical supervision. It is therefore proposed to develop and build such a system and to conduct extended home based trials in three people with tetraplegia.

ELIGIBILITY:
Inclusion Criteria:

* Have a spinal cord injury that has resulted in tetraplegia affecting hand function.
* Minimal spasticity of wrist muscle.
* Able to do shoulder elevation.
* Upper limb passive range of motion should be within normal limit.
* Age group: 18 years and above.
* Able to understand and comply with assessment procedures.
* Able to give informed consent.
* Able to produce a muscle contraction using electrical stimulation in sufficient muscles produce a functional grip.

Exclusion Criteria:

* Using a cardiac pacemaker, defibrillator or other sensitive implanted device.
* Pregnant or planning to become pregnant over the course of the study.
* A history of poorly controlled epilepsy.
* If there is malignancy on the hand or arm.
* If younger than 18
* Severe contracture of wrist and finger joints.
* Painful shoulder.
* Suffering from significant autonomic dysreflexia in response to FES.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Grasp Release Test (GRT) | Start of study - 30 minutes building up to 60 minutes over a four week period
  Test to be completed both with and without the device - exercise daily for 30 minutes, building up to 60 minutes over a four week period
Grasp Release Test (GRT) | At the end of the clinical phase (week 10) - 30 minutes building up to 60 minutes over a four week period
  Test to be completed both with and without the device - exercise daily for 30 minutes, building up to 60 minutes over a four week period
Grasp Release Test (GRT) | At the end of the home phase for participants taking the device home (week 18) - 30 minutes building up to 60 minutes over a four week period
  Test to be completed both with and without the device - exercise daily for 30 minutes, building up to 60 minutes over a four week period

SECONDARY OUTCOMES:
Measurement of palmar grip | At the start of the study - 30 minutes
  Test to be completed both with and without the device
Measurement of pinch grip | At the start of the study - 30 minutes
  Test to be completed both with and without the device
Measurement of palmar grip | At the end of the clinical phase (week 10) - 30 minutes
  Test to be completed both with and without the device
Measurement of pinch grip | At the end of the clinical phase (week 10) - 30 minutes
  Test to be completed both with and without the device
Measurement of palmar grip | At the end of the home phase for participants taking the device home (week 18) - 30 minutes
  Test to be completed both with and without the device
Measurement of pinch grip | At the end of the home phase for participants taking the device home (week 18) - 30 minutes
  Test to be completed both with and without the device

OTHER OUTCOMES:
Two Point Discrimination Test | At the start of the study
  Test to be completed both with and without the device
Two Point Discrimination Test | At the end of the clinical phase (week 10)
  Test to be completed both with and without the device
Two Point Discrimination Test | At the end of the home phase for participants taking the device home (week 18)
  Test to be completed both with and without the device

CONTACTS AND LOCATIONS:
Overall Officials: Ian Swain, Professor, Study Director — Professor in Technology & Design; Paul Taylor, Professor, Principal Investigator — Consultant Clinical Scientist - Salisbury District Hospital
Locations (1):
- Salisbury District Hospital, Salisbury, Wiltshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided